CLINICAL TRIAL: NCT03607604
Title: Application of UCPCR as a Testing Tool for Identification of MODY Patients in the UAE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC018
Record Dates: First submitted 2018-06-26; First posted 2018-07-31 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Maturity-onset Diabetes of the Young
Keywords: MODY; Diabetes Mellitus; UCPCR; Monogenic Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Mason-Type Diabetes; Diabetes Mellitus | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA will be extracted from collected blood samples for genetic analysis (suspected MODY cases)

GROUPS / COHORTS (3):
- Autoantibody Negative: Patients who are autoantibody negative (could potentially be either MODY or type 2 diabetes patients)
  Suspected MODY patients will be candidates for next generation sequencing (NGS)
  Interventions: Genetic: Next generation sequencing (NGS)
- Diabetes Mellitus, Type 1: Patients diagnosed with type 1 diabetes mellitus
  Patients with positive UCPCR and negative autoantibodies results will be suspected with MODY and will be candidates for next generation sequencing (NGS)
  Interventions: Genetic: Next generation sequencing (NGS)
- Non Diabetic: Individuals not diagnosed with any type of diabetes (but could be diagnosed with IFG and/or IGT)

INTERVENTIONS:
Genetic: Next generation sequencing (NGS) — Patients will be tested for known MODY genes with specific focus on HNF1A, GCK and HNF4A genes. Furthermore, gene panel testing may be performed for any known diabetes genes.If the results are negative, WES/WGS will be performed in patients suspected of having MODY for identification of novel MODY mutations.
  Other Names: NGS panel; Whole exome/genome sequencing (WES/WGS)
  Groups: Autoantibody Negative; Diabetes Mellitus, Type 1

SUMMARY:
The study aims to investigate the validity of 2 hour post-prandial UCPCR test in paediatric and adult patients with diabetes duration greater than 2 and 5 years, respectively, for the purposes of distinguishing between patients with type 1 diabetes and MODY in the UAE population.

DETAILED DESCRIPTION:
Urinary C-peptide creatinine ratio (UCPCR) is a non invasive measure of endogenous insulin secretion and has been shown to be effective in identifying Maturity Onset Diabetes of the Young (MODY) from Type 1 Diabetes in adults and paediatric population. Here in the UAE, diabetes prevalence is at 18.9% of the general population and patients are medically treated according to their diabetes type. Currently identification of patients with MODY poses multiple challenges and in some instances results in wrongful diagnosis and treatment of the patients. Most commonly, patients are treated as having type 1 diabetes and given unnecessary insulin injections.

Making correct diabetes diagnosis is pivotal for appropriate disease management. Currently, a set of criteria including age of onset of diabetes (<30 years), BMI<25kg/m2 and absence of islet-cell and GAD auto-antibodies are applied in order to identify potential Maturity Onset Diabetes of the Young (MODY) patients. This has to be followed by genetic testing before final diagnosis is made. Although the set criteria increase the probability of identifying MODY patients, fully discriminating between MODY and type 1 diabetes can still be difficult. As such, some MODY patients (e.g. with mutations in HNF1A or HNF4A genes) are wrongfully treated with insulin when sulphonylureas would be efficient enough for management of their diabetes.

This study will consists of three groups; patients who are autoantibody negative (divided into patients with potential MODY and patients with type 2 diabetes), patients diagnosed with type 1 diabetes and patients who do not have diabetes at the time of recruitment (selected randomly and will include patients with other diagnoses such as IFG and/or IGT). All groups will consist of paediatric patients (≤18 years of age) and adult patients (age of onset of diabetes ≤ 30 years).

The scientific aims of the study are:

* Validating UCPCR as an in-house test that can potentially be used for clinical purposes.
* Measuring UCPCR in the study cohort and testing if a cutoff of 0.7nmol/mmol in children and 0.2nmol/mmol in adults will apply to population of interest (ie UAE population).
* Using operating characteristic curves to identify the optimal UCPCR cut-off for discriminating diabetes subtypes in.
* Confirming the UCPCR results through genetic analysis of the samples.
* Validating positive genetic test results by performing mutational analysis on the parents of the patient.
* Potentially identifying novel MODY mutations in the study population.
* conducting UCPCR measurements for patients who have been clinically and genetically diagnosed with MODY. This will assist the investigators in confirming the cutoff values for MODY diagnosis.
* Successfully estimating the background prevalence of MODY in diabetes patients in the Emirates of Abu Dhabi.

ELIGIBILITY:
Inclusion Criteria:

* patients with age and age of diabetes onset of <18 years
* patients with age of ≥18 years and age of diabetes onset of ≤30 years

Exclusion Criteria:

- patients with age of ≥18 years and age of diabetes onset of >30 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending Imperial College London Diabetes Centre, UAE.
Sampling Method: Non-Probability Sample
Enrollment: 778 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary C-peptide Creatinine Ratio (UCPCR) | 2 hours post-prandial
  Measuring UCPCR in our study cohort and testing if a cutoff of 0.7nmol/mmol in children and 0.2nmol/mmol in adults will apply to our population of interest (ie UAE population).

SECONDARY OUTCOMES:
Receiver operating characteristic (ROC) curve | through study completion, an average of 1 year
  Using receiver operating characteristic (ROC) curves to identify the optimal UCPCR cut-off for discriminating diabetes subtypes in our study population.
Genetic analysis | through study completion, an average of 2 year
  Confirming our UCPCR results through genetic analysis of the samples.
Positive genetic result analysis | through study completion, an average of 2 year
  Validating positive genetic test results by performing mutational analysis on the parents of the patient.
Novel MODY genes and mutations | through study completion, an average of 2 year
  Identifying novel MODY genes and/or mutations in the study population through next generation sequencing methodologies
UCPCR measurements | through study completion, an average of 2 year
  Conducting UCPCR measurements for patients who have been clinically and genetically diagnosed with MODY. This will assist us in confirming the cutoff values for MODY diagnosis.
Prevalence of MODY | through study completion, an average of 2 year
  Estimating the background prevalence of MODY in diabetes patients in the Emirates of Abu Dhabi.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Lessan, MBBS FRCP MD, Principal Investigator — Imperial College London Diabetes Centre
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates